CLINICAL TRIAL: NCT03555240
Title: Regional Registry-based Biobank Development and Pharmacogenetic Analysis: Synergistic Strategies Driving Towards Personalized Medicine in Rheumatoid Arthritis Management
Brief Title: Regional Registry-based Biobank Development and Pharmacogenetic Analysis in Rheumatoid Arthritis
Acronym: RABiobank
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Regione Emilia Romagna - Italy within PRU-Liberati project (Unknown)
Responsible Party: Sponsor
Other Study IDs: PRUA1GR-2013-00000203
Record Dates: First submitted 2018-05-18; First posted 2018-06-13 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2018-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with Rheumatoid Arthritis: Patient with Rheumatoid Arthritis living in the Emilia Romagna Italian region whom samples will be collected for the Biobank creation and Pharmacogenetic analysis
  Interventions: Other: Biobank creation and Pharmacogenetic analysis

INTERVENTIONS:
Other: Biobank creation and Pharmacogenetic analysis — Collection of biological samples (blood, serum, plasma) form patient enrolled in the Emilia Romagna rheumatoid arthritis registry and genotyping genomic DNA samples, and assessing the association between genotypes and response to biological drugs, using multivariate and data-mining approaches that includes also clinical and demographic parameters.

SUMMARY:
Aim of this project is the building-up of an integrated model of multidisciplinary research tools to support large-scale and high-quality disease-based studies.

DETAILED DESCRIPTION:
Biologics have revolutionized rheumatoid arthritis (RA) management, with a great impact on patient that justifies treatment with these high-cost drugs. Nevertheless, timing and proper therapeutic decision making remain the main challenge in clinical practice.

Pharmacogenetics approach might open promising perspectives, increasing our understanding on genetic-related drug efficacy. Nevertheless, to ensure feasibility and reliability of translational applications of this strategy in clinical practice, large population-based research studies represent a crucial key step.

Objectives

Major aim of this project is the building-up of an integrated model of multidisciplinary research tools to support large-scale and high-quality disease-based studies. The main targets of this proposal will be:

* to develop a disease-based biobank, integrated with already established Emilia-Romagna regional RA Registry, providing a large-scale prospective collection and storing of multiple biological samples
* to perform a pharmacogenetic study analyzing a panel of gene variants potentially influencing the response to Tumor Necrosis Factor (TNF) blockers. Methods
* Biobank development. A step-wise plan will be considered for: designing biobank governance frame-work, defining Standard Operating Procedures, implementing information system resources. All these procedures will be applied for collecting, processing and storing biological samples of patients included in regional RA registry.
* Pharmacogenetic study. A panel of candidate gene variants will be studied in genomic DNA from 300 patients enrolled in the regional RA registry. The association between genotypes and response to biological drugs will be assessed by data-mining approach, and a predictive model will be defined. Expected Results This proposal will create a disease-based biobank, tightly integrated with the already established Emilia-Romagna regional RA Registry, and pave the way towards personalized therapy applications in Rheumatology.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Arthritis Rheumatoid according American College of Rheumatology (ACR)1987 or according ACR/European League Against Rheumatism (EULAR) 2010 criteria
2. Patients with new diagnosis or patients already diagnosed with active disease [with Disease Activity Score (DAS) 28 > o = 4,2] or patients switching therapy
3. Male and female patients of minimum 18 years old
4. Provision of informed consent

Exclusion Criteria:

1) Patients living outside Emilia Romagna region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with residents in Emilia Romagna Region, partecipating to the regional rheumatoid arthritis registy
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2014-10-27 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Biobank creation | through study completion, an average of 5 years
  Collection of biological samples from patients included into Emilia Romagna Rheumatoid Arthritis Registry

SECONDARY OUTCOMES:
Identification of genes potentially predictive of response to biological drugs | at 12 Months
  Pharmacogenetics analysis of genes involved in the response to biological drugs

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Assirelli, BSc, Principal Investigator — Rizzoli Orthopedic Institute
Locations (10):
- Italy (10):
  - Rheumatology Unit IRCCS Orthopedic Rizzoli Institute, Bologna, BO
  - Rheumatology Unit, Internal Medicine Department of Internal Medicine and Nephrology diseases and Aging, Bologna, BO
  - Rheumatology Unit, Department of Internal Medicine Buflini Hospital, Cesena, FC
  - Medical Genetics Unit, Dept. of Biomedical and Specialty Surgery, Ferrara, FE
  - Rheumatology Unit S.Anna University Hospital, Ferrara, FE
  - Rheumatology Unit, Internal Medicine Department Morgagni Hospital, Forlì, Fo
  - Unit of Internal Medicine, Medical Internistic Department Ospedale Santa maria delle croci, Ravenna, RA
  - Division of Rheumatology Azienda Ospedaliera-IRCC S, Reggio Emilia, Reggio Emilia, RE
  - Department of Internal Medicine Infermis' Hospital, Rimini, RN
  - Laboratory of Immunorheumatology and Tissue Regeneration IRCC Rizzoli Orthopedic Institute, Bologna

IPD SHARING:
Plan to Share IPD: No
No Plan

REFERENCES:
- [Background] Boonen A, Severens JL. The burden of illness of rheumatoid arthritis. Clin Rheumatol. 2011 Mar;30 Suppl 1:S3-8. doi: 10.1007/s10067-010-1634-9. Epub 2011 Feb 26. PMID 21359507
- [Background] Hamilton SR, Chatrian GE, Mills RP, Kalina RE, Bird TD. Cone dysfunction in a subgroup of patients with autosomal dominant cerebellar ataxia. Arch Ophthalmol. 1990 Apr;108(4):551-6. doi: 10.1001/archopht.1990.01070060099057. PMID 2322158
- [Background] Scott DL. Biologics-based therapy for the treatment of rheumatoid arthritis. Clin Pharmacol Ther. 2012 Jan;91(1):30-43. doi: 10.1038/clpt.2011.278. Epub 2011 Dec 14. PMID 22166850
- [Background] Ruderman EM. Overview of safety of non-biologic and biologic DMARDs. Rheumatology (Oxford). 2012 Dec;51 Suppl 6:vi37-43. doi: 10.1093/rheumatology/kes283. PMID 23221586
- [Background] Prajapati R, Plant D, Barton A. Genetic and genomic predictors of anti-TNF response. Pharmacogenomics. 2011 Nov;12(11):1571-85. doi: 10.2217/pgs.11.114. PMID 22044414

DOCUMENTS (1):
  • Study Protocol (2014-05-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT03555240/Prot_000.pdf